CLINICAL TRIAL: NCT06017544
Title: Glucagon-like Peptide-1 Receptor Agonists (GLP-1RAs) and Sodium-glucose Cotransporter-2 Inhibitors (SGLT2is) Combination Therapy and Major Adverse Cardiovascular Events After Acute Myocardial Infarction: an Observational Study in Patients with Type 2 Diabetes.
Brief Title: GLP-1RAs) and SGLT2is Combination Therapy and MACEs in Patients with Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, Professor of Medicine, University of Campania Luigi Vanvitelli
Other Study IDs: 0124.082023
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2; Myocardial Infarction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- T2DM patients with GLP-1 RA: T2DM patients hospitalized due to AMI as a primary diagnosis, both STEMI and NSTEMI, referred for PCI, and under GLP-1 RA.
  Interventions: Procedure: PCI
- T2DM patients with SGLT2-is: T2DM patients hospitalized due to AMI as a primary diagnosis, both STEMI and NSTEMI, referred for PCI, and under SGLT2-is.
  Interventions: Procedure: PCI
- T2DM patients with GLP-1 RA plus SGLT2-is: T2DM patients hospitalized due to AMI as a primary diagnosis, both STEMI and NSTEMI, referred for PCI, and under GLP-1 RA plus SGLT2-is.

INTERVENTIONS:
Procedure: PCI — The T2DM affected by AMI will be referred for receiving PCI.
  Groups: T2DM patients with GLP-1 RA; T2DM patients with SGLT2-is

SUMMARY:
Management of type 2 diabetes mellitus (T2DM) has evolved from a glucocentric to a cardiometabolic approach. Both glucagon-like peptide-1 receptor agonists (GLP-1RAs) and sodium-glucose cotransporter-2 inhibitors (SGLT2is) reduce cardiovascular and kidney outcomes in T2DM patients with a low hypoglycemia risk. The T2DM di per se still carries a higher risk of mortality and major cardiovascular complications, doubling the case fatality rate. Tacking that GLP-1RAs and SGLT2is have different mechanisms of action, resulting in complementary pharmacokinetics and pharmacodynamics, the combination use may present clinical efficacy and safety in T2DM patients with AMI. However, there is limited clinical evidence that supports the combined use of these drugs, and there are currently no studies investigating the effects of combination treatment in T2DM patients with acute cardiovascular events, on MACE as well as on myocardial post-infarction rescue. Therefore, authors will conduct an observational prospective study to evaluate the effects GLP-1RAs and SGLT2is combination therapy on MACE such as mortality, acute coronary syndrome and heart failure, and myocardial salvage index (MSI) after acute myocardial infarction (AMI) in T2DM patients.

DETAILED DESCRIPTION:
Management of type 2 diabetes mellitus (T2DM) has evolved from a glucocentric to a cardiometabolic approach. Consequently, choosing anti-hyperglycemic therapies with proven cardiovascular and renal benefits is now a cornerstone of T2DM management. Both glucagon-like peptide-1 receptor agonists (GLP-1RAs) and sodium-glucose cotransporter-2 inhibitors (SGLT2is) individually been shown to reduce cardiovascular and kidney outcomes in T2DM patients with a low hypoglycemia risk. Thus, the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD) indifferently recommended both classes as first-line therapy in patients with T2DM and established atherosclerotic cardiovascular disease (ASCVD) or multiple ASCVD risk factors to reduce the risk of major adverse cardiovascular events (MACE). However, although these drugs have singularly improved survival in both T2DM and non-T2DM patients with acute myocardial infarction (AMI), the presence of T2DM still carries a higher risk of mortality and major cardiovascular complications, doubling the case fatality rate. Tacking that GLP-1RAs and SGLT2is have different mechanisms of action, resulting in complementary pharmacokinetics and pharmacodynamics, the combination use may present clinical efficacy and safety in T2DM patients with AMI. In such patients, the ADA-EASD 2022 consensus report also recommends the combination of GLP-1RAs and SGLT2is when the haemoglobin A1c (HbA1c) target is not reached with a drug from one of the two classes [6]. However, there is limited clinical evidence that supports the combined use of these drugs, and there are currently no studies investigating the effects of combination treatment in T2DM patients with acute cardiovascular events, on MACE as well as on myocardial post-infarction rescue. Therefore, authors will conduct an observational prospective study to evaluate the effects GLP-1RAs and SGLT2is combination therapy on MACE such as mortality, acute coronary syndrome and heart failure, and myocardial salvage index (MSI) after acute myocardial infarction (AMI) in T2DM patients.

Methods Study design Authors will perform a three-centres, prospective observational study with post-enrollment allocation of groups. Consecutive T2DM patients, treated with GLP-1 RA or SGLT-2i, with acute myocardial infarction will be enlisted for this study. All T2DM patients hospitalized due to AMI as a primary diagnosis, both ST-elevation myocardial infarction (STEMI) and non-ST-elevation myocardial infarction (NSTEMI), referred for percutaneous coronary intervention (PCI), will be initially screened from January 1, 2018, through December 31, 2022. Patients will be stratified according to their glycemic control at the time of hospitalization. As suggested by the ADA Standard of Care in diabetes, T2DM patients with HbA1c <7% wil be considered in good glycemic control. T2DM patients in good glycemic control will be further stratified according to GLP-1 RA or SGLT-2i treatment for at least 3 months before index hospitalization. According to the ADA and the EASD recommendations, the combination of GLP-1RA and SGLT2i will be adopted in T2DM in poor glycemic control (HbA1c >7%). Exclusion criteria will include evidence of heart failure, valvular defects, malignant neoplasms, or secondary causes of hypertension. After discharge from the hospital, all T2DM patients will be managed and followed quarterly for two years after PCI as outpatients to maintain HbA1c level at <7%, blood glucose level of 80-130 mg/dl, and post-prandial blood glucose level of <180 mg/dl. A multifactorial person-centered approach will be adopted during the follow-up to maintain the glycemic, weight, and cardiorenal goals. According to the ADA and EASD recommendations, patients initially treated with GLP-1 RA or SGLT-2i will be switched to combination therapy when HbA1c was >7% during follow-up. The myocardial rescue will be evaluated by MSI (SPECT) before the hospital discharge and at the end of follow-up, as previously described. Briefly, authors will use the total perfusion deficit (TPD) to calculate the area at risk (AAR) and infarct size. Regarding quantitative gated SPECT (QGS) data, QGS software (Cedars-Sinai Medical Center, Los Angeles, CA, USA) will be used to calculate LV function and volume. The SPECT data will be collected and calculated as follows: AAR (%) as TPD on 123I-BMIPP polar-map; infarct size (%) as TPD on 99mTc-tetrofosmin polar-map; MSI = (AAR - infarct size)/AAR; LV volume and function (LV end-systolic volume [LVESV], LV end-diastolic volume [LVEDV], and LV ejection fraction [LVEF]) based on 99mTc-tetrofosmin QGS data. All SPECT analyses will be performed by experienced radiology technologists who will be unaware of patients' and angiographic characteristics With regard to full medical therapy, the protocol stated that the use of concomitant treatment should be as uniform as possible and according to evidence-based international guidelines for AMI. Patients with incomplete data or lost during follow-up will be excluded from the analysis.

Study endpoints The study's primary endpoint will be the composite of mortality, acute heart failure, and acute coronary syndrome (SCA) requiring hospitalization. To avoid interference, each patient could only account for one event classification. The secondary endpoint will be the MSI.

Statistical analysis Data will be presented as numbers and frequencies for categorical variables and as means and standard deviations for continuous variables. The distribution of variables will be assessed with the Shapiro-Wilk test. The differences between the three study groups will be assessed using ANOVA and Mann-Whitney tests, as appropriate. Categorical variables will be described using frequencies and percentages and compared using χ2 -test. Differences among the three groups for continuous and categorical variables will be assessed by ANOVA and χ2-test, respectively. Cox regression analysis will be used to examine the association between the combination of GLP-1RAs and SGLT2is and the incidence of the composite outcome and will be adjusted for age, sex, BMI, diabetes duration, 24-months HbA1c mean levels, admission HbA1c mean levels 3-months HbA1c mean levels, LDL-cholesterol, troponin, creatinine, the prevalence of hypertension, dyslipidemia and smoking. P values < 0.05 will be considered statistically significant. All calculations will be performed using SPSS 29.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive T2DM patients, treated with GLP-1 RA or SGLT-2i, with AMI;
* both STEMI and NSTEMI patients referred for PCI;

Exclusion criteria:

* heart failure and valvular defects;
* inflammatory chronic diseases;
* neoplastic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM patients, treated with GLP-1 RA or SGLT-2i, hospitalized due to AMI (STEMI and NSTEMI), and referred for PCI. The patients will be stratified according to their glycemic control at the time of hospitalization: T2DM patients with HbA1c <7% will be considered in good glycemic control.
  T2DM patients in good glycemic control will be further stratified according to GLP-1 RA or SGLT-2i treatment for at least 3 months before index hospitalization. The combination of GLP-1RA and SGLT2i will be adopted in T2DM in poor glycemic control (HbA1c >7%). After discharge from the hospital, all T2DM patients will be managed and followed quarterly for two years after PCI as outpatients to maintain HbA1c level at <7%, blood glucose level of 80-130 mg/dl, and post-prandial blood glucose level of <180 mg/dl.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
MACE | 12 months
  The study's primary endpoint was the composite of mortality, acute heart failure, and acute coronary syndrome (SCA) requiring hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Celestino Sardu, Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marfella R, Prattichizzo F, Sardu C, Rambaldi PF, Fumagalli C, Marfella LV, La Grotta R, Frige C, Pellegrini V, D'Andrea D, Cesaro A, Calabro P, Pizzi C, Antonicelli R, Ceriello A, Mauro C, Paolisso G. GLP-1 receptor agonists-SGLT-2 inhibitors combination therapy and cardiovascular events after acute myocardial infarction: an observational study in patients with type 2 diabetes. Cardiovasc Diabetol. 2024 Jan 6;23(1):10. doi: 10.1186/s12933-023-02118-6. PMID 38184582